CLINICAL TRIAL: NCT06137144
Title: A Modular Phase I/II, Open-label, Multicentre Study to Evaluate the Safety, Tolerability, and Efficacy of AZD3470, a PRMT5 Inhibitor, as Monotherapy and in Combination With Anticancer Agent(s) in Participants With Relapsed/Refractory Haematologic Malignancies
Brief Title: AZD3470 as Monotherapy and in Combination With Anticancer Agents in Participants With Relapsed/Refractory Haematologic Malignancies.
Acronym: PRIMAVERA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D9971C00001; 2023-506747-42-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-11-02; First posted 2023-11-18 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Lymphoma; Non-Hodgkin; Hodgkin Lymphoma
Keywords: Haematologic Malignancies; Hodgkin lymphoma; MTAP deficient; PRMT5
MeSH Terms: conditions — Lymphoma; Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Module 1: Part A (Dose Escalation) and Part B (Dose Expansion/Optimization) (Experimental): In Part A, participants with Relapsed/Refractory classical Hodgkin Lymphoma (cHL) will take AZD3470 tablets orally until PD, unacceptable toxicity, or withdrawal of consent.
  In Part B, adult and adolescent participants with r/r cHL will take AZD3470 tablets orally until PD, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: AZD3470

INTERVENTIONS:
Drug: AZD3470 — AZD3470 is a novel, potent and selective, second-generation, Methylthioadenosine (MTA)-selective, small molecule inhibitor of PRMT5.

SUMMARY:
This study is designed to evaluate the safety, tolerability, PK and preliminary efficacy following oral administration of AZD3470 as a monotherapy, and in combination with other anticancer agents in participants with haematologic malignancies.

DETAILED DESCRIPTION:
This is a FTiH modular, Phase I/II, open-label, multicentre, dose escalation and expansion study in participants with r/r haematologic malignancies. The study is designed to evaluate the safety, tolerability, PK and preliminary efficacy following oral administration of AZD3470 as a monotherapy, and in combination with other anticancer agents in participants with haematologic malignancies.

This study will follow a modular protocol design evaluating AZD3470 as monotherapy and in combination with other anticancer agents. New cohorts (including further monotherapy expansion) and new modules for combination treatments may be added as protocol amendments in the future based on emerging supportive preclinical and/or clinical data.

Module 1 Part A includes a dose escalation of AZD3470 monotherapy in participants with r/r haematologic malignancies, initially focused on r/r cHL. Dose escalation cohorts will evaluate the safety, tolerability, PK, and preliminary efficacy in participants with r/r cHL.

Module 1 Part B optimization/expansion cohorts may be opened at selected dose levels. These cohorts will further characterise the safety, PK, and preliminary efficacy of AZD3470 to support dose optimization. Both adult and adolescent participants with r/r cHL will be eligible for this part of the study. Adolescent participants will only be enrolled once there is sufficient PK and safety data in adults. A preliminary effect of food on AZD3470 pharmacokinetics will be explored in this part of the study.

The protocol may be amended in the future to incorporate further expansion of cHL at the RP2D, additional monotherapy cohorts in other hematologic malignancies, and/or additional modules investigating AZD3470 in combination with other anticancer agents.

ELIGIBILITY:
Inclusion criteria

* Adequate organ and bone marrow function.
* In Part A (dose escalation), participants must be aged ≥ 18 years at the time of signing the informed consent. In Part B (dose optimization/expansion), participants must be at least 15 years of age.
* Histologically confirmed documented diagnosis of r/r cHL based on criteria established by the World Health Organization
* Must provide FFPE baseline tumour tissue to meet the minimum tissue requirement for central MTAP expression determination.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Contraceptive use by males or females should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Module 1 (cHL):

* At least 1 radiographically measurable, and/or FDG-avid lymphoma lesion > 1.5 cm.
* Participants must have documented r/r active disease, must have previously received at least 3 prior lines of therapy (including Brentuximab Vedotin and anti-PD-1 therapy) for the treatment of cHL, and must have exhausted all available therapies with demonstrated clinical benefit.

Exclusion criteria

* Any significant laboratory finding or any severe and uncontrolled medical condition.
* Active CNS involvement by lymphoma, leptomeningeal disease, or spinal cord compression.
* Serologic active HBV or HCV infection.
* Known to have tested positive for HIV.
* Active gastrointestinal disease or other condition that will interfere with oral therapy.
* Any of the following cardiac criteria:

  * Mean resting QTcF > 470 msec or clinically important abnormalities in rhythm (ventricular arrhythmias and uncontrolled atrial fibrillation)
  * Factors that increase the risk of QTc prolongation or risk of arrhythmic events
  * Cardiac procedures or conditions within the last 6 months: Coronary artery bypass graft (CABG), percutaneous coronary intervention (PCI) or heart valve intervention vascular stent implantation, acute coronary syndrome / myocardial infarction, uncontrolled angina pectoris, use of therapeutic anti-coagulation for treatment of active thromboembolic events.
  * Severe valvular heart disease
  * Congestive heart failure Grade II to Grade IV
  * Prior or current cardiomyopathy
  * Uncontrolled hypertension
  * Brain perfusion problems such as haemorrhagic or thrombotic stroke (including transient ischemic attacks)
* Unresolved non-haematological toxicities of Grade > 1 from prior anticancer therapy (excluding peripheral neuropathy, vitiligo, alopecia, and endocrine disorders that are controlled with replacement hormone therapy, and asymptomatic laboratory abnormalities), unless immune-mediated.
* History of another primary malignancy.
* History of significant haemoptysis or haemorrhage within 4 weeks of the first dose of study treatment.
* Requires ongoing immunosuppressive therapy, including systemic corticosteroids.
* Prior treatment with a MAT2A inhibitor or a PRMT5 inhibitor.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2026-05-08 (Estimated); Study Completion 2026-05-08 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | From Screening until 28 days after the last dose of study medication.
  AEs: Number of patients with adverse events by system organ class and preferred term.
  SAEs: Number of patients with serious adverse events by system organ class and preferred term.
Incidence of DLTs (Dose Escalation only) | From first dose of AZD3470 to end of Cycle 1 (each cycle is 21 days).
  In the Dose Escalation cohorts in Part A, the number of participants with at least 1 dose-limiting toxicity (DLT), which is any toxicity defined as a DLT in the Clinical Study Protocol.

SECONDARY OUTCOMES:
Part A and Part B: Response endpoints - Objective Response Rate (ORR)/Complete Response Rate (CRR) | From first dose (Cycle 1 Day 1, each cycle is 21 days) until disease progression or the last evaluable assessment in the absence of progression (assessed approximately up to 2 years).
  ORR is defined as the proportion of participants who have a CR or PR and CRR is defined as the proportion of participants who have a CR.
  Assessment of ORR/CRR will be done according to the Lugano Classification for cHL.
Part A and Part B: Response endpoints - Duration of Response (DoR) | From first dose (Cycle 1 Day 1, each cycle is 21 days) until disease progression or death, whichever comes first (assessed approximately up to 2 years).
  The time from the date of first documented response until the date of documented progression as assessed by the investigator according to the Lugano classification for cHL, or death due to any cause.
Part A and Part B: Progression-free Survival (PFS) | Non-randomized study parts: from first dose (each cycle is 21 days) until disease progression or death, whichever comes first. Randomized parts: from date of randomization until disease progression or death, whichever comes first (approx up to 2 years).
  Time from date of first dose (non- randomised study parts) or date of randomization (randomised study parts) until progression as assessed by the investigator according to the Lugano Classification for cHL, or death due to any cause.
Part A and Part B: Overall Survival (OS) | Non-randomized study parts: From first dose (Cycle 1 Day 1, each cycle is 21 days) until death. Randomized study parts: from date of randomization until the date of death due to any cause (assessed approximately up to 2 years).
  Time from date of first dose (non-randomised study parts) or date of randomization (randomised study parts) until the date of death due to any cause.
Part A and Part B: Maximum observed plasma drug concentration (Cmax) | From Cycle 1 Day 1 (each cycle is 21 days) to EoT, at predefined intervals throughout the treatment period (for each patient this is expected to be approximately 6 months).
  Assessed to characterize the plasma PK profile of AZD3470.
Part A: Dose normalised maximum observed plasma drug concentration (Cmax) | From Cycle 1 Day 1 (each cycle is 21 days) to EoT, at predefined intervals throughout the treatment period (for each patient this is expected to be approximately 6 months).
  Assessed to characterize the plasma PK profile of AZD3470.
Part A: Accumulation ratio for maximum observed plasma drug concentration (Cmax) | From Cycle 1 Day 1 (each cycle is 21 days) to EoT, at predefined intervals throughout the treatment period (for each patient this is expected to be approximately 6 months).
  Assessed to characterize the plasma PK profile of AZD3470.
Part A and Part B: Minimum observed plasma drug concentration (Cmin) | From Cycle 1 Day 1 (each cycle is 21 days) to EoT, at predefined intervals throughout the treatment period (for each patient this is expected to be approximately 6 months).
  Assessed to characterize the plasma PK profile of AZD3470.
Part A and Part B: Time to reach peak or maximum observed concentration following drug administration (Tmax) | From Cycle 1 Day 1 (each cycle is 21 days) to EoT, at predefined intervals throughout the treatment period (for each patient this is expected to be approximately 6 months).
  Assessed to characterize the plasma PK profile of AZD3470.
Part A and Part B: Area under the plasma concentration-curve over the dosing interval (AUCtau) | From Cycle 1 Day 1 (each cycle is 21 days) to EoT, at predefined intervals throughout the treatment period (for each patient this is expected to be approximately 6 months).
  Assessed to characterize the plasma PK profile of AZD3470.
Part A: Dose normalized area under the plasma concentration-curve over the dosing interval (AUCtau) | From Cycle 1 Day 1 (each cycle is 21 days) to EoT, at predefined intervals throughout the treatment period (for each patient this is expected to be approximately 6 months).
  Assessed to characterize the plasma PK profile of AZD3470.
Part A: Accumulation ratio for area under the plasma concentration-curve over the dosing interval (AUCtau) | From Cycle 1 Day 1 (each cycle is 21 days) to EoT, at predefined intervals throughout the treatment period (for each patient this is expected to be approximately 6 months).
  Assessed to characterize the plasma PK profile of AZD3470.
Part A: Cumulative amount (%) of drug recovered unchanged in urine during dosing interval (Ae,tau) | From Cycle 1 Day 1 to end of Cycle 1 at predefined intervals throughout the cycle (each cycle is 21 days).
  Assessed to characterize the urine PK profile of AZD3470.
Part A: Renal clearance (Clr) | From Cycle 1 Day 1 to end of Cycle 1 at predefined intervals throughout the cycle (each cycle is 21 days).
  Assessed to characterize the urine PK profile of AZD3470.
Part B: Ratio of maximum observed plasma drug concentration (Cmax) under fed/fasted state | From Cycle 1 Day 1 to Cycle 2 Day 1 at predefined intervals (each cycle is 21 days).
  Preliminary food effect on plasma PK of AZD3470 administered as a monotherapy in participants enrolled in dose expansion.
Part B: Time to reach peak or maximum observed concentration following drug administration (Tmax) under fed conditions | From Cycle 1 Day 1 to Cycle 2 Day 1 at predefined intervals (each cycle is 21 days).
  Preliminary food effect on plasma PK of AZD3470 administered as a monotherapy in participants enrolled in dose expansion.
Part B: Time to reach peak or maximum observed concentration following drug administration (Tmax) under fasted conditions | From Cycle 1 Day 1 to Cycle 2 Day 1 at predefined intervals (each cycle is 21 days).
  Preliminary food effect on plasma PK of AZD3470 administered as a monotherapy in participants enrolled in dose expansion.
Part B: Ratio of area under the plasma concentration-curve over the dosing interval (AUCtau) under fed/fasted state | From Cycle 1 Day 1 to Cycle 2 Day 1 at predefined intervals (each cycle is 21 days).
  Preliminary food effect on plasma PK of AZD3470 administered as a monotherapy in participants enrolled in dose expansion.

CONTACTS AND LOCATIONS:
Locations (19):
- United States (5):
  - Research Site, Miami, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Boston, Massachusetts
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Houston, Texas
- Research Site, Nedlands, Australia
- France (4):
  - Research Site, Créteil
  - Research Site, Lille
  - Research Site, Pierre-Bénite
  - Research Site, Villejuif
- Research Site, Cologne, Germany
- Italy (3):
  - Research Site, Alessandria
  - Research Site, Bologna
  - Research Site, Milan
- Research Site, Seoul, South Korea
- Spain (2):
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
- United Kingdom (2):
  - Research Site, Manchester
  - Research Site, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patientlevel data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home